CLINICAL TRIAL: NCT01907997
Title: Effects of Systemic Lidocaine on Postoperative Quality of Recovery After Robot-assisted Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0342
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Thyroid Cancer
Keywords: Systemic lidocaine, Intravenous lidocaine infusion, postoperative pain, quality of recovery, Robot-assisted thyroidectomy, thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Experimental): Intravenous lidocaine infusion group
  Interventions: Drug: Systemic intravenous lidocaine infusion
- Group C (Placebo Comparator): Intravenous normal saline infusion - control group
  Interventions: Drug: normal saline infusion

INTERVENTIONS:
Drug: Systemic intravenous lidocaine infusion — In group L, intravenous lidocaine infusion(0.1mg/kg) for 10minutes after induction of anesthesia. After 10 minutes, lidocaine infusion continued at rate of 3mg/kg/hr during operation, and discontinued before move the patients to PACU.
  Arms: Group L
Drug: normal saline infusion — In group C, the patients receive same volume of normal saline
  Arms: Group C

SUMMARY:
Systemic lidocaine infusion may improve the patients' recovery quality and chronic post surgical pain after robot-assisted thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-65
* ASA class I and II
* Thyroid cancer patients who are scheduled for elective robot-assisted thyroidectomy

Exclusion Criteria:

* Allergy to local anesthetics or contraindication to use of lidocaine
* Pregnancy
* Severe cardiovascular disease
* Renal failure
* Liver failure
* Neurologic and psychologic disease
* Chronic treatment with analgesics

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 40(QoR-40) score | 24hours after operation day
  Assessing change of the Quality of recovery 40(QoR-40) score between 24hours before and after operation

SECONDARY OUTCOMES:
Assessing the presence of chronic postsurgical pain(CPSP) | 24hours after operation day
aspect and site of CPSP | 24hours after operation day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei universiy college of medicine, Seoul, South Korea

REFERENCES:
- [Derived] Choi KW, Nam KH, Lee JR, Chung WY, Kang SW, Joe YE, Lee JH. The Effects of Intravenous Lidocaine Infusions on the Quality of Recovery and Chronic Pain After Robotic Thyroidectomy: A Randomized, Double-Blinded, Controlled Study. World J Surg. 2017 May;41(5):1305-1312. doi: 10.1007/s00268-016-3842-1. PMID 27896411